CLINICAL TRIAL: NCT03929692
Title: Effect of a Cardiovascular Health Promotion Program in Youth - The Tyrolean Early Vascular Ageing-study
Acronym: EVA-Tyrol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Collaborators: Tiroler Landeskrankenanstalten GmbH (TILAK) (Unknown); Tiroler Gebietskrankenkasse (TGKK) (Unknown); InfPro IT Solutions GmbH (Unknown); Genossenschaft Milchhof Sterzing (Dairy Farm Sterzing) (Unknown); Austrian Research Promotion Agency FFG (K Project) (Unknown); Public Health Service of South Tyrol, Italy (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EVA1
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Atherosclerosis; Life Style
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Intervention Model Description: The Intervention Group (mean age 15-16 years at the baseline and 17-18 years at follow-up) will be compared to a Control Group (mean age 17-18 years) that did not participate in the health promotion program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Other): Intervention will consist of (1) enhancing knowledge about CVDs, (2) individual medical counseling based on the results of the baseline examination, (3) providing an online health promotion tool and (4) involvement of participants in planning and conduction of health promotion projects.
  Interventions: Behavioral: Multi-layer health promotion program; Other: Standard health education
- Control Group (Other): Adolescents of same age as intervention group at follow-up examination that did not participate in health promotion program.
  Interventions: Other: Standard health education

INTERVENTIONS:
Behavioral: Multi-layer health promotion program
  Arms: Intervention Group
Other: Standard health education

SUMMARY:
Atherosclerosis - the main cause of cardiovascular diseases - starts already in childhood. The Tyrolean Early Vascular Ageing-study aims to improve the vascular health of Tyrolean adolescents by a multi-layer intervention program.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVDs) are the leading non-communicable cause of death. Primary prevention measures aim to improve the awareness of the individual risk profile and promote healthy lifestyle. Multiple evaluations have shown, that atherosclerosis - the main cause of CVDs - begins already early in life. Therefore, prevention programs have to start already in childhood.

The EVA-Tyrol study is a prospective, biomedical cohort study. 2000 participants will be recruited from high schools and training companies spread over North- and East-Tyrol (Austria) and South-Tyrol (Italy). For the 1500 participants included in the intervention group two examinations will be scheduled within a two-year interval. Participants will be in the 10th grade (mean age, 15-16 years) at the baseline and in the 12th grade (mean age, 17-18 years) at the follow-up examination. 500 participants in the 12th grade without participation in a health promotion program will serve as a control group. The 2000 participants equal roughly 5% of the Tyrolean population of the included age-group. Medical examination includes an extensive questionnaire, anthropometric measurements, fasting blood sampling, high-resolution ultrasound of the common carotid artery, and carotid-femoral pulse wave velocity. Active intervention will consist of (1) enhancing knowledge about CVDs, (2) individual medical counseling based on the results of the baseline examination, (3) providing an online health promotion tool and (4) involvement of participants in planning and conduction of health promotion projects. Main outcome parameter is the difference in the number of ideal health metrics as defined by the American Heart Association between the intervention and control group.

This study aims to improve cardiovascular health in Tyrolean adolescents and to evaluate the efficacy of this multi-layer health promotion program. Moreover, the investigators expect numerous insights in the prevalence of vascular risk conditions and early vascular pathologies in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Intervention group: Participants must be in 10th school grade or aged 15 to 16 years when recruited in training companies.
* Control Group: Participants must be in 12th school grade or aged 17 to 18 years when recruited in training companies.

Exclusion Criteria:

- none

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2102 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Effect of health promotion. | 2 years
  Difference in the number of AHA's seven health goals in the ideal range between the intervention and the control Group.

SECONDARY OUTCOMES:
Change in vascular health. | 2 years
  Difference (decrease, stagnation, increase) of the number of achieved number of AHA's seven health goals in the ideal range between the baseline and the follow-up examination of the intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Kiechl-Kohlendorfer, MD, Principal Investigator — Medical University of Innsbruck; Michael Knoflach, MD, Principal Investigator — Medical University of Innsbruck
Locations (2):
- Department of Pediatrics II (Neonatology), Medical University of Innsbruck, Innsbruck, Tyrol, Austria
- Department of Pediatrics, Bruneck Hospital, Bruneck, Trentino-Alto Adige, Italy

IPD SHARING:
Plan to Share IPD: No
Anonymized data can be shared in academic cooperations. Request for data can be addressed to the principal investigators with an appropriate research question.

REFERENCES:
- [Derived] Winder B, Zollner-Kiechl S, Bernar B, Gande N, Staudt A, Stock AK, Hochmayr C, Geiger R, Griesmacher A, Kiechl S, Kiechl-Kohlendorfer U, Knoflach M; Early Vascular Ageing (EVA)-Tyrol Study Group. The association of physical activity and carotid intima-media-thickness in adolescents-data of the prospective early vascular ageing-tyrol cohort study. Front Pediatr. 2025 Feb 6;13:1527132. doi: 10.3389/fped.2025.1527132. eCollection 2025. PMID 39981205
- [Derived] Bernar B, Gande N, Stock AK, Staudt A, Pechlaner R, Hochmayr C, Kaltseis K, Winder B, Zollner-Kiechl S, Broessner G, Geiger R, Kiechl S; Early Vascular Ageing (EVA) Tyrol Study Group; Kiechl-Kohlendorfer U, Knoflach M. Early Vascular Ageing in adolescents with migraine with aura: a community-based study. BMC Cardiovasc Disord. 2023 Aug 1;23(1):384. doi: 10.1186/s12872-023-03409-2. PMID 37528337
- [Derived] Hochmayr C, Ndayisaba JP, Gande N, Staudt A, Bernar B, Stock K, Zollner-Kiechl S, Geiger R, Griesmaier E, Knoflach M, Kiechl-Kohlendorfer U; Early Vascular Ageing (EVA) Study Group. Cardiovascular health profiles in adolescents being born term or preterm-results from the EVA-Tyrol study. BMC Cardiovasc Disord. 2023 Jul 25;23(1):371. doi: 10.1186/s12872-023-03360-2. PMID 37488472
- [Derived] Kaltseis K, Frank F, Bernar B, Zollner-Kiechl S, Winder B, Kiechl-Kohlendorfer U, Knoflach M, Broessner G; Early Vascular Ageing (EVA) Tyrol Study Group. Primary headache disorders in adolescents in North- and South-Tyrol: Findings of the EVA-Tyrol-Study. Cephalalgia. 2022 Sep;42(10):993-1004. doi: 10.1177/03331024221088997. Epub 2022 Mar 25. PMID 35331020
- [Derived] Winder B, Kiechl SJ, Gruber NM, Bernar B, Gande N, Staudt A, Stock K, Hochmayr C, Geiger R, Griesmacher A, Anliker M, Kiechl S, Kiechl-Kohlendorfer U, Knoflach M; Early Vascular Ageing (EVA)-Tyrol Study Group. The association of allergic asthma and carotid intima-media thickness in adolescence: data of the prospective early vascular ageing (EVA)-Tyrol cohort study. BMC Cardiovasc Disord. 2022 Jan 18;22(1):11. doi: 10.1186/s12872-021-02452-1. PMID 35042472
- [Derived] Kiechl SJ, Staudt A, Stock K, Gande N, Bernar B, Hochmayr C, Winder B, Geiger R, Griesmacher A, Anliker M, Kiechl S, Kiechl-Kohlendorfer U, Knoflach M, Pechlaner R; Early Vascular Ageing (EVA) Study Group *. Predictors of Carotid Intima-Media Thickness Progression in Adolescents-The EVA-Tyrol Study. J Am Heart Assoc. 2021 Sep 21;10(18):e020233. doi: 10.1161/JAHA.120.020233. Epub 2021 Sep 6. PMID 34482715
- [Derived] Gande N, Pechlaner R, Bernar B, Staudt A, Stock K, Hochmayr C, Geiger R, Kiechl-Kohlendorfer U, Knoflach M; Early Vascular Aging (EVA) Study Group. Cardiovascular health behaviors and associations of sex, age, and education in adolescents - Results from the EVA Tyrol study. Nutr Metab Cardiovasc Dis. 2021 Apr 9;31(4):1286-1292. doi: 10.1016/j.numecd.2020.11.002. Epub 2020 Nov 10. PMID 33558093
- [Derived] Bernar B, Gande N, Stock KA, Staudt A, Pechlaner R, Geiger R, Griesmacher A, Kiechl S, Knoflach M, Kiechl-Kohlendorfer U; Early Vascular Aging (EVA) Study Group. The Tyrolean early vascular ageing-study (EVA-Tyrol): study protocol for a non-randomized controlled trial : Effect of a cardiovascular health promotion program in youth, a prospective cohort study. BMC Cardiovasc Disord. 2020 Feb 5;20(1):59. doi: 10.1186/s12872-020-01357-9. PMID 32024473